CLINICAL TRIAL: NCT02120807
Title: A Phase I Trial of Certolizumab in Combination With Chemotherapy for Patients With Stage IV Lung Adenocarcinomas
Brief Title: Certolizumab in Combination With Chemotherapy for Patients With Stage IV Lung Adenocarcinomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-063
Record Dates: First submitted 2014-04-21; First posted 2014-04-23 (Estimated); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Stage IV Lung Adenocarcinoma
Keywords: Certolizumab; Cisplatin; Pemetrexed; thoracic; 13-063
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Certolizumab Pegol; Cisplatin; Pemetrexed

ARMS (1):
- certolizumab, cisplatin and pemetrexed (Experimental): Patients will receive certolizumab with 6 cycles of cisplatin & pemetrexed. Cycle of chemo will be 3 weeks. Certolizumab will be adm in the following fashion: first dose administered at the time of treatment initiation, second dose will be given after 2 weeks of treatment, third dose after four weeks of treatment, & subsequent doses given every 4 weeks thereafter. Patients will be monitored for progression of disease using RECIST 1.1 with scans to be performed every 6 weeks. Posttreatment biopsies will be performed at the time of treatment discontinuation. Two dose levels of certolizumab will be tested, 200mg & 400mg. A non-therapeutic cohort of 10 patients with adenocarcinomas who will be undergoing standard of care treatment with platinum based chemotherapy + pemetrexed +/- bevacizumab will be consented for blood draws before each cycle of treatment. This blood will be analyzed for cytokines and will serve as a reference for the experimental arm.
  Interventions: Drug: Certolizumab; Drug: cisplatin; Drug: pemetrexed

INTERVENTIONS:
Drug: Certolizumab
Drug: cisplatin
Drug: pemetrexed

SUMMARY:
The purpose of this study is to test the safety of certolizumab when it is given with the chemotherapy drugs cisplatin and pemetrexed. Cisplatin and pemetrexed are two chemotherapy drugs used in the treatment of lung cancer. The investigators want to find out what effects, good and/or bad, certolizumab has on the patient and lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated stage IV lung adenocarcinoma confirmed at MSKCC
* Age 18 years or older
* Karnofsky Performance Status ≥ 70
* Patients with locally treated, stable, and/or asymptomatic brain metastases are eligible.
* Adequate bone marrow, liver and renal function, as specified below:
* Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L
* Hemoglobin ≥ 8 g/dL
* Platelets ≥ 100 x 109/L
* Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN) (except for patients with documented Gilbert's Syndrome)
* AST and ALT ≤ 2.5 x ULN or ≤ 5 x ULN if liver metastases are present
* Serum creatinine ≤ 1.5 x upper limit of normal or creatinine clearance ≥ 60ml/min for patients with creatinine levels above institutional normal.
* Negative PPD test
* For women of child-bearing potential, negative pregnancy test within 14 days prior to starting treatment
* Men and women of childbearing age must be willing to use effective contraception while on treatment and for at least 3 months thereafter
* Presence of at least one site of measurable disease as defined by the Response Evaluation Criteria in Solid Tumors
* Archival tissue (10 Unstained Slides - 5 micron sections) from a core biopsy performed and received within 30 days before signing consent or ability to have a fresh core biopsy performed
* Biopsy cannot be from any cytology or bone specimen
* Biopsy site must be amenable to re-biopsy at the end of the study
* Ability to provide written, informed consent

Exclusion Criteria:

* Hypersensitivity to platinum agents
* Ongoing use of investigational agents or use of investigational agents within the last four weeks
* Prior use of agents for TNF-alpha blockade
* History of rheumatoid arthritis, inflammatory bowel disease, or psoriatic arthritis
* Baseline hearing deficit (CTCAE version 4.0 grade 2 or higher)
* Ongoing bacterial, viral, or antifungal infection requiring antimicrobial treatment with the exception of thrush
* Active tuberculosis or untreated, latent tuberculosis

  o If a patient has signs, symptoms, or a history suggestive of active tuberculosis, evaluation by an infectious disease physician will be required and active tuberculosis ruled-out prior to enrollment.
* Acute or chronic Hepatitis B or C infection
* Known HIV infection requiring antiretroviral medications and those with AIDS
* Active herpes zoster infection
* Non-healed infected skin ulcers
* History of myocardial infarction or unstable angina within the past 12 months
* Ongoing use of other immunosuppressive medications, including oral steroids and excluding topical steroids
* Women who are breastfeeding Prior history of other malignancy with the exclusion of localized prostate cancer, non-melanomatous skin cancer, ductal carcinoma or lobular carcinoma in situ of the breast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04-15 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated does (MTD) | 2 years
  A standard 3+3 dose-escalation scheme will be used to test two doses of certolizumab: dose level A (200mg) and dose level B (400mg), in combination with the standard dose of chemotherapy. In addition, two de-escalation doses are planned, if dose level A proves too toxic: dose level C (chemotherapy at 75% of the standard dose + certolizumab 200mg) and dose level D (chemotherapy at 75% of the standard dose + certolizumab 400mg)..The MTD is the highest dose at which ≤ 1/6 patients experiences a DLT. Please see the dose escalation schema for exact dose level details.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 2 years
  Patients will be followed from the first drug administration until disease progression (by RECIST 1.1) or death, whichever comes first. Patients alive who have not progressed by the end of the study time will be censored at the time of the last available follow-up. PFS probability will be estimated using Kaplan-Meier methods.
Immunohistochemical staining | 2 years
  Biopsies will be performed pre- and post-treatment in all patients and will undergo immunohistochemical staining of TNF-alpha, CXCL1/2, and S100A8/9. Staining will be scored from 0-4. The difference in IHC score from post-treatment to baseline will be compared between patients who have, at minimum, evidence of stable disease during treatment (CR+PR+SD) and the remaining patients, using non-parametric Wilcoxon signed rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Paik, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering West Harrison, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memorial Sloan Kettering Cancer Center at Phelps Memorial Hospital Center, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/